CLINICAL TRIAL: NCT07124728
Title: Impact of Syntrillo's Telehealth Service on Stroke Risk Factor Reduction in At-risk Patients
Brief Title: Syntrillo Telehealth Stroke Risk Reduction Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Syntrillo, Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025003
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Hypertension (HTN); Stroke Prevention; Cardiovascular Risk Factor
Keywords: stroke prevention; telehealth; telemedicine; blood pressure; remote patient monitoring; digital health; heart rate variability; inflammation; hypertension
MeSH Terms: conditions — Hypertension; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telemedicine Stroke Prevention Program (Experimental): Participants will receive a 6-month personalized telehealth intervention including remote patient monitoring, blood pressure management, lifestyle counseling, wearable monitoring, and multidisciplinary telemedicine visits via the Healthie platform.
  Interventions: Behavioral: Technology-enabled Telehealth Care Plan; Device: Blood Pressure Monitoring Device; Device: Tenovi Smart Pillbox; Device: Wearable Activity Trackers (Fitbit or Apple Watch); Other: Healthie EHR; Other: Secure Messaging Platforms (TigerConnect, Weave, AirCall); Drug: Antihypertensive Medication Management; Drug: Statin Medication Management; Drug: Antiplatelet or Anticoagulant Therapy; Procedure: Laboratory Blood Test Collection

INTERVENTIONS:
Behavioral: Technology-enabled Telehealth Care Plan — Participants receive a 6 month personalized telehealth intervention via a multidisciplinary care team, delivering care via a secure digital platform, including education, risk assessment, lifestyle coaching, medical history review, and stroke risk reduction planning. The Healthie EHR is used for communication, documentation, and data integration. Syntrillo Navigators and neurology providers conduct onboarding, telemedicine visits, and coordination with patient's primary care providers and care team.
Device: Blood Pressure Monitoring Device — Participants will receive a cellular-enabled, FDA-cleared blood pressure monitor supplied by Tenovi. Blood pressure is measured twice daily during baseline and at least once daily throughout the 6-month intervention. Data is transmitted via a secure gateway to the Healthie EHR for real-time monitoring and analysis.
Device: Tenovi Smart Pillbox — Participants receive a connected 7-day smart pillbox that detects compartment openings and refills. Medication adherence data is uploaded in real time to a secure dashboard and integrated into the EHR.
Device: Wearable Activity Trackers (Fitbit or Apple Watch) — Participants will utilize a commercially available wearable activity tracker to monitor step counts, resting heart rate, and heart rate variability. This data is integrated into the EHR. Devices will be provided if participants do not already own one.
Other: Healthie EHR — HIPAA-compliant electronic medical record system used for participant management, secure communication, clinical documentation, and device data integration, consisting of custom workflows used for risk tracking and care planning.
Other: Secure Messaging Platforms (TigerConnect, Weave, AirCall) — Participants and providers may communicate using secure messaging platforms for appointment reminders, assessments, and care support, to enhance participation engagement and care coordination.
Drug: Antihypertensive Medication Management — Participants may be prescribed or have existing antihypertensive regimens adjusted (ACE inhibitors, beta blockers, calcium channel blockers, diuretics, etc) by neurologists or nurse practitioners based on individual risk assessments and clinical findings during the study. Changed will be recorded in EHR.
Drug: Statin Medication Management — Lipid-lowering medications, including statins, may be initiated or adjusted as part of participants' care plans. Medication use is guided by cardiovascular risk and AHA guidelines. Changed will be recorded in EHR.
Drug: Antiplatelet or Anticoagulant Therapy — Participants with atrial fibrillation or elevated cardiovascular risk may be started on or have changes to antiplatelet or anticoagulant therapy. Medication decisions are made by neurologist or nurse practitioners during telemedicine visits. Changed will be recorded in EHR.
Procedure: Laboratory Blood Test Collection — Blood samples may be collected at baseline and at 6 months to assess inflammation through high-sensitivity C-reactive protein.

SUMMARY:
A prospective, single-arm, open-label study evaluating the impact of Syntrillo's telehealth program on stroke risk factors, particularly blood pressure, among 68 high-risk patients. The 6-month intervention includes personalized remote care with blood pressure monitoring, wearable tracking, and multidisciplinary telehealth visits.

DETAILED DESCRIPTION:
Participants ≥30 years old with hypertension and at least one of the following conditions: atrial fibrillation, diabetes, chronic kidney disease (stage 2 or higher), obesity (class 2 or higher), obstructive sleep apnea, coronary artery disease, hyperlipidemia, carotid stenosis (of 50% or greater), and/or congestive heart failure will be enrolled in a 6-month telehealth intervention focused on stroke risk reduction. The program includes use of home blood pressure monitors, smart pillboxes, wearable activity trackers, and a multidisciplinary team for personalized care. Primary endpoint is change in systolic blood pressure. Additional endpoints include diastolic BP, inflammatory markers (hs-CRP), and cardiovascular biomarkers (resting heart rate, HRV). The study is single-arm, non-randomized, and exploratory in design.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 30
* Diagnosis of hypertension
* One or more of the following:
* Dtrial fibrillation
* Diabetes
* Chronic kidney disease (stage 2+)
* Obesity (class 2+)
* Obstructive sleep apnea
* Coronary artery disease
* Hyperlipidemia
* Carotid stenosis (greater than or equal to 50%)
* Congestive heart failure

Exclusion Criteria:

* History of stroke or TIA
* Inability to consent or understand study
* Residence in long-term acute care facility
* Inability to ambulate independently
* Non-English speaking
* No internet access
* Not residing in Virginia
* Pregnancy or suspected pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure | Baseline to 6 months
  This measure evaluates the average change in systolic blood pressure (SBP), which is the pressure in the arteries when the heart beats. Blood pressure is measured by participants at home using a Tenovi FDA-cleared digital blood pressure monitor. Baseline SBP is calculated using the first 10 valid readings taken during the initial week of monitoring. The 6-month value is calculated from the last 10 valid readings taken in the final week of the intervention. The study aims to observe a reduction of at least 10 mmHg in average SBP over the intervention period.

SECONDARY OUTCOMES:
Change in Diastolic Blood Pressure | Baseline to 6 months
  This measure evaluates the average change in systolic blood pressure (SBP), which is the pressure in the arteries when the heart beats. Blood pressure is measured by participants at home using a Tenovi FDA-cleared digital blood pressure monitor. Baseline SBP is calculated using the first 10 valid readings taken during the initial week of monitoring. The 6-month value is calculated from the last 10 valid readings taken in the final week of the intervention. The study aims to observe a reduction of at least 10 mmHg in average SBP over the intervention period.
Change in Systolic Blood Pressure Variability | Baseline to 6 months
  This measure assesses the variability of systolic blood pressure (SBP) as measured by the standard deviation (SD) of SBP readings. Variability is calculated from 20 readings collected at baseline (first 2 weeks) and another 20 readings at the end of the intervention (final 2 weeks). Measurements are taken using the Tenovi home blood pressure monitor. The target is a 10% reduction in the standard deviation of SBP values, indicating more stable blood pressure control.
Change in Pulse Pressure | Baseline to 6 months
  This measure evaluates the change in pulse pressure (PP), defined as the difference between systolic and diastolic blood pressure. PP is a marker of arterial stiffness and cardiovascular risk. It is calculated from 20 home blood pressure readings collected at the start and again at the end of the 6-month intervention. Measurements are obtained using the Tenovi device. The study target is a reduction of at least 5 mmHg in average pulse pressure.
Change in High-Sensitivity C-Reactive Protein (hs-CRP) | Baseline to 6 months
  This measure examines changes in high-sensitivity C-reactive protein (hs-CRP), a blood marker of systemic inflammation and cardiovascular risk. hs-CRP levels are measured from blood samples collected at baseline and again at the 6-month time point. The study aims to observe a mean reduction of at least 20% in hs-CRP concentration over the course of the intervention.
Change in Resting Heart Rate | Baseline to 6 months
  This measure evaluates the change in resting heart rate (RHR), defined as the number of heartbeats per minute when the body is at rest. RHR is measured using participant-worn Fitbit or Apple Watch devices. The average RHR is calculated from 20 data points collected during the initial monitoring period and compared with 20 data points collected in the final weeks of the intervention. The study aims to observe a mean decrease of at least 5 beats per minute in resting heart rate.
Change in Heart Rate Variability | Baseline to 6 months
  This measure tracks changes in heart rate variability (HRV), a measure of autonomic nervous system function. HRV is assessed using the standard deviation of NN intervals (SDNN), collected from data provided by Fitbit or Apple Watch wearable devices. Baseline SDNN is calculated from 40 measurements during the first 2 weeks, and compared to 40 measurements taken during the final 2 weeks of the study. The target is a 10% or greater increase in average SDNN over the study period.

IPD SHARING:
Plan to Share IPD: No
De-identified data may be used internally for algorithm development and clinical workflow optimization, but will not be publicly shared.